CLINICAL TRIAL: NCT01482533
Title: Tissue Culture Versus Swab Culture in Prosthetic Joint Infections
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Rothman Institute Orthopaedics (Other)
Responsible Party: Principal Investigator, Tiffany Morrison, MS, Manager, Clinical Trials, Rothman Institute Orthopaedics
Other Study IDs: RIUJPar01-2011
Record Dates: First submitted 2011-11-28; First posted 2011-11-30 (Estimated); Last update posted 2011-11-30 (Estimated); Status verified 2011-11

CONDITIONS: Revision Total Hip Arthroplasty; Revision Total Knee Arthroplasty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Revision Total Hip Arthroplasty
- Revision Total Knee Arthroplasty

SUMMARY:
The main purpose of this study is to compare the effectiveness and accuracy of tissue cultures and swab cultures to diagnose prosthetic joint infection.

ELIGIBILITY:
Inclusion Criteria:

1. Patients are scheduled for revision TJA surgery.
2. Subjects are willing to sign the informed consent document.

Exclusion Criteria:

1. Subject not willing to sign the informed consent document.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients undergoing revision surgery for an infection in their knee or hip components.
Sampling Method: Non-Probability Sample

CONTACTS AND LOCATIONS:
Locations (1):
- Rothman Institute, Philadelphia, Pennsylvania, United States